CLINICAL TRIAL: NCT00521079
Title: EMPOWER Clinical Trial: Vagal Blocking for Obesity Control
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D00343-000
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Excess weight loss; Vagus nerve; Vagal blocking; vBloc(TM) therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vBloc (Experimental): Subjects implanted with a functional Maestro System device that delivers therapy (Therapy ON).
  Interventions: Device: Therapy ON
- Placebo (Sham Comparator): Subjects implanted with a functional Maestro System device that does NOT deliver therapy (Therapy OFF).
  Interventions: Device: Therapy OFF

INTERVENTIONS:
Device: Therapy ON — Intermittent, programmable, intra-abdominal vagal blocking device that delivers therapy (Therapy ON)
  Other Names: Maestro System
  Arms: vBloc
Device: Therapy OFF — Active intra-abdominal placebo device that delivers no therapy (Therapy OFF)
  Other Names: Maestro System
  Arms: Placebo

SUMMARY:
This is a randomized multi-center study being done to measure the ability of a new medical device, Maestro System, to safely reduce body weight over five years in people who are considered obese.

DETAILED DESCRIPTION:
The Maestro System is a neuromodulation system that consists of implantable and external components.

Implantable components: two leads (one electrode each for the anterior and posterior intra-abdominal vagal nerve trunks) that are connected to an implantable neuroregulator.

External components: one programmable, battery-powered, ambulatory external controller connected via a small, flexible cable to a cutaneous transmit coil that is positioned externally over the neuroregulator. A clinician programmer that transmits information to the controller and uploads data from the controller.

All non-diabetic subjects will be randomized in a 2:1 allocation to therapy ON or therapy OFF groups. All type 2 diabetes mellitus subjects will be randomized in a 1:1 allocation to therapy ON or therapy OFF groups.

All subjects will receive blinded therapy through the 12-month follow-up visit. All subjects will participate in a medical weight management program.

ELIGIBILITY:
Inclusion criteria

1. Informed consent.
2. Body mass index (BMI) ≥ 40 kg/m2 to 45 kg/m2 or BMI ≥ 35 kg/m2 to 39.9 kg/m2 with one or more obesity related co-morbid condition. Co-morbid conditions may include one or more of the following:

   * Type 2 diabetes mellitus (note: type 2 diabetics are allowed at selected centers only, see Inclusion criterion #5)
   * Hypertension as defined by systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg a) treated or untreated with systolic ≥140 mmHg or diastolic ≥90 mmHg or b) treated with systolic <140 mmHg and diastolic <90 mmHg
   * Dyslipidemia as defined by total cholesterol ≥200 or LDL ≥130 a) treated or untreated with total cholesterol ≥200 or LDL ≥130 or b) treated with total cholesterol <200 or LDL <130
   * Sleep apnea syndrome (confirmed by overnight p02 studies)
   * Obesity related cardiomyopathy
3. Females or males Note: females of child-bearing potential must have a negative urine pregnancy test at Screen and also within 14 days of implant procedure followed by physician-approved contraceptive regimen for the duration of the study period.
4. 18-65 years of age inclusive.
5. Type 2 diabetes mellitus subjects (at selected centers, limited to approximately 34 subjects) with:

   * Glycosylated hemoglobin (Hb A1c) 6.5 - 9 % inclusive at screening visit.
   * Onset: 10 years or less since initial diagnosis.
   * Stable treatment regimen: no change in oral hypoglycemic treatment regimen within past 3 months.
   * Currently not using insulin therapy, GLP-1 receptor agonists (e.g., exenatide), or DPP-4 inhibitors (e.g., sitagliptin) for diabetes treatment and have not been on these treatments in the past 6 months.
   * Creatinine within normal reference range.
   * No history of proliferative retinopathy.
   * No history of peripheral neuropathy.
   * No history of autonomic neuropathy.
   * No history of coronary artery disease, with or without angina pectoris.
   * No history of peripheral vascular disease.
6. Failure to respond to supervised diet/exercise program(s) in which the subject was engaged for at least 6 months within the last five years.
7. Ability to complete all study visits and procedures.

Exclusion criteria

1. Concurrent chronic pancreatic disease.
2. History of Crohn's disease and/or ulcerative colitis.
3. History of bariatric surgery, fundoplication, gastric resection or major upper-abdominal surgery (acceptable surgeries include cholecystectomy, hysterectomy).
4. History of pulmonary embolism or blood coagulation disorders.
5. Clinically significant hiatal hernias known from subject's medical record as or determined by upper endoscopy prior to implant if they have not had one done during the previous 6 months that specifically reported on the presence or absence of hiatal hernia making reference to the Z-line and/or diaphragmatic notch, in order to rule out subjects with hiatal hernia that may require surgical repair (to support exclusion criterion #7).
6. Current portal hypertension and/or esophageal varices.
7. Intra-operative exclusion: hiatal hernia requiring surgical repair or extensive dissection at esophagogastric junction at time of surgery.
8. Treatment with weight-loss prescription drug therapy within the prior three months and the use of prescription drug therapy or the use over-the-counter weight loss preparations for the duration of the trial.
9. Smoking cessation within the prior six months.
10. Known genetic cause of obesity (e.g., Prader-Willi Syndrome).
11. Overall sustained reduction of more than 10% of body weight in the previous 12 months.
12. Physician-prescribed pre-operative diet with intent to lose weight prior to surgery (note: a) study subject may continue any personal diet they were on prior to study enrollment [see exclusion criterion #24] b) standardized EMPOWER weight management program to be initiated in all subjects at time of activation, approximately two weeks after implant)
13. Current type 1 diabetes mellitus (DM).
14. Current or recent history (within 12 months) of ongoing bulimia.
15. Current alterations in treatment for thyroid disorders (stable treatment regimen for prior three months acceptable).
16. Current alterations in treatment for epilepsy (stable treatment regimen for prior six months acceptable).
17. Current treatment for peptic ulcer disease (previous history acceptable).
18. Chronic (more than 4 weeks of daily use) treatment with narcotic analgesic drug regimens (treatment with non-steroidal anti-inflammatory drugs acceptable).
19. Current alterations in treatment regimens of anti-cholinergic drugs, including tricyclic antidepressants (stable treatment regimen for prior six months acceptable).
20. Current medical condition that, in the opinion of the investigator, would make subject unfit for surgery under general anesthesia or that would be exacerbated by intentional weight loss. Some examples include diagnosis of cancer, recent heart attack, recent stroke or recent serious trauma.
21. Presence of permanently implanted electrical powered medical device or implanted gastrointestinal device or prosthesis (e.g., pacemakers, implanted defibrillators, neurostimulators etc.).
22. Planned or contemplated use of Magnetic Resonance Imaging (MRI) or oncological radiation during the course of the trial.
23. Significant psychiatric disorders that, in the opinion of the investigator, may interfere with subject's ability to follow study procedures and/or instructions.
24. Current, active member of an organized weight loss program (e.g., Weight Watchers, TOPS).
25. Current participant in another weight loss study or other clinical trials.
26. Have a friend or family member who is currently participating or is planning to participate in this clinical trial.
27. Patient reported:

    * inability to walk for about 10 minutes without stopping,
    * feeling of pain in chest when doing physical activity,
    * feeling of pain in chest when not doing physical activity. Note: unless pain in chest in known to be related to upper gastrointestinal disorders such as gastroesophageal reflux disease or heartburn.
28. Clinically significant cardiac rhythm disorder that requires either medical and/or surgical intervention (e.g., paroxysmal or chronic atrial fibrillation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Billington, MD, Principal Investigator — VA Medical Center, Minneapolis, MN / University of Minnesota; Michael Sarr, MD, Principal Investigator — Mayo Clinic
Locations (15):
- United States (13):
  - HonorHealth (formerly Scottsdale Bariatric Center), Scottsdale, Arizona
  - Scripps Clinic, La Jolla, California
  - University of California, Irvine Medical Center, Orange, California
  - Stanford University Medical Center, Stanford, California
  - Cleveland Clinic - Florida, Weston, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic - Ohio, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Institute of Weight Control, Sydney, New South Wales
  - Adelaide Bariatric Center - Flinders Private Hospital, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | vBloc | Placebo
Started | 192 | 102
Surgical Roll-In | 9 | 5
Completed | 178 | 97
Not Completed | 14 | 5
Not completed — Adverse Event | 7 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | vBloc | Placebo | Total
Number analyzed (Participants) | 183 | 97 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 97 | 280
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (9.7) | 45.6 (10.6) | 45.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 83 | 248
  Male | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  United States | 142 | 77 | 219
  Australia | 41 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Excess Weight Loss (EWL) With the Maestro System
Description: Observe at least a 10% greater percentage excess weight loss (%EWL) with vBloc therapy delivered by the Maestro System compared to sham 12 months following randomization using MetLife Method (ideal body weight is calculated based on Metropolitan Height and Weight Tables)
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Error); unit: Percentage of excess weight loss
Arm/Group | vBloc | Placebo
Number analyzed (Participants) | 165 | 88
Percentage of excess weight loss | 17 (2) | 16 (2)

2. Primary Outcome: Rate of System and Procedure-related Serious Adverse Events (SAEs).
Description: To estimate the rate of serious, system- and procedure-related adverse events associated with the Maestro System.
Time Frame: 1 Year
Measure: Number; unit: Events
Arm/Group | vBloc | Placebo
Number analyzed (Participants) | 192 | 102
Events | 6 | 3

3. Secondary Outcome: Percentage of Participants Achieving 25% Excess Weight Loss (%EWL)
Description: To evaluate the percentage of participants achieving 25% excess weight loss from baseline (implant) to 12 months between treatment groups.
Time Frame: Baseline and 1 Year
Measure: Number; unit: Percentage of subjects
Arm/Group | vBloc | Placebo
Number analyzed (Participants) | 183 | 97
Percentage of subjects | 22 | 25

ADVERSE EVENTS:
Description: Includes roll-in subjects.
Groups:
- Placebo: Subjects implanted with a functional Maestro System device that does NOT delivers therapy (Therapy OFF).
Arm/Group | vBloc | Placebo
Serious Adverse Events (participants affected / at risk) | 23/192 | 12/102
Other Adverse Events (participants affected / at risk) | 146/192 | 70/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vBloc (N=192) | Placebo (N=102)
Incision pain incision site (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection neuroregulator site (Infections and infestations) | 2 (2) | 1 (1)
Lead impedance high (Surgical and medical procedures) | 0 (0) | 1 (1)
Neuroregulator malfunction (Surgical and medical procedures) | 1 (1) | 0 (0)
Pain abdominal (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pain neuroregulator site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Bleeding other (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cardiac abnormality (Cardiac disorders) | 1 (1) | 0 (0)
Cold/flu/respiratory tract infection (General disorders) | 1 (1) | 0 (0)
Gallbladder disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Infection other (Infections and infestations) | 1 (1) | 1 (1)
Large bowel dysfunction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (General disorders) | 8 (8) | 6 (6)
Pain other (General disorders) | 1 (1) | 0 (0)
Reaction to medicines (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vBloc (N=192) | Placebo (N=102)
Bloating Abdominal (Gastrointestinal disorders) | 10 (10) | 7 (8)
Chest Pain (General disorders) | 19 (19) | 2 (2) — Primarily related to the sensation of therapy. Generally occurred early with mild to moderate severity.
Constipation (Gastrointestinal disorders) | 32 (38) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 23 (29) | 15 (20)
Eructation (Gastrointestinal disorders) | 20 (22) | 10 (11)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 47 (57) | 15 (17)
Incision pain incision site (Surgical and medical procedures) | 7 (7) | 8 (8)
Nausea (Gastrointestinal disorders) | 32 (40) | 9 (9)
Pain Abdominal (Gastrointestinal disorders) | 32 (38) | 19 (22)
Pain neuroregulator site (Skin and subcutaneous tissue disorders) | 42 (47) | 28 (30)
Skin reaction to coil/coil adhesion method (General disorders) | 18 (21) | 8 (9)
Wound redness or irritation (Skin and subcutaneous tissue disorders) | 11 (12) | 4 (5)
Cold/flu/respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 93 (170) | 46 (101)
Depression (Psychiatric disorders) | 24 (24) | 6 (6)
Energy decreased (General disorders) | 14 (15) | 3 (3)
Headache (General disorders) | 20 (22) | 6 (7)
Edema (Cardiac disorders) | 9 (9) | 3 (3)
Emesis (vomiting) (Gastrointestinal disorders) | 20 (20) | 8 (10)
Out of range lab values (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Vitamin or mineral insufficiency (Metabolism and nutrition disorders) | 14 (18) | 6 (8)
Cramps abdominal (Gastrointestinal disorders) | 8 (8) | 6 (7)
Reaction to medicines (General disorders) | 9 (10) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 14 (15) | 9 (13)
Anxiety (Psychiatric disorders) | 5 (7) | 5 (5)
Trauma (Musculoskeletal and connective tissue disorders) | 8 (11) | 9 (12)
Paresthesia (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
Two confounding efficacy factors: Variable hours of therapy in both arms due to inconsistent external power source use and altered vagal excitability in the control arm due to small electrical inputs delivered to vagal nerves for safety checks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less